CLINICAL TRIAL: NCT00576056
Title: Phase II Trial of Transcatheter Arterial Chemoembolization (TACE) Plus Oral Sorafenib (BAY 43-9006, Nexavar®) for Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Effectiveness and Safety Study of TACE Plus Oral Sorafenib for Unresectable HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Bayer Healthcare is no supplying the study drug
Sponsor: University of Pittsburgh (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Susan Lamson, RN, BA, RN BA, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-047
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular; Carcinoma; TACE; Sorafenib; Transcatheter Arterial Chemoembolization; Nexavar; Unresectable
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tace and Sorafenib (Experimental): Patients with unresectable HCC will be treated with TACE in combination with oral sorafenib administration. TACE will be accomplished with gelatin microspheres (Embospheres) following delivery of 125 mg/m2 of cisplatin. Oral sorafenib (400 mg BID) will start the next day after the first TACE treatment.
  Interventions: Drug: Sorafenib; Drug: TACE

INTERVENTIONS:
Drug: Sorafenib — Oral sorafenib (400 mg BID) will start the next day after the first TACE treatment until unacceptable toxicity occurs, or until study termination.
  Other Names: Nexavar
Drug: TACE — TACE will be accomplished with gelatin microspheres (Embospheres) following delivery of 125 mg/m2 of cisplatin.
  Other Names: Transarterial Chemoembolization

SUMMARY:
The purpose of this study is to determine if TACE plus Sorafenib will improve outcome in patients with advanced hepatocellular carcinoma (HCC) not amenable to surgery.

DETAILED DESCRIPTION:
The proposed study will make an important contribution to understanding not only the safety and efficacy of sorafenib in addition to TACE in patients diagnosed with unresectable HCC, but this will also be the first clinical trial with sorafenib to assess the effects of this novel therapy on HRQL. Understanding the effects of sorafenib on HRQL is critical in the treatment of HCC secondary to the modest benefits in survival that have been reported with conventional therapies. Our team has one of the largest experiences in evaluating HRQL in patients diagnosed with unresectable hepatocellular carcinoma. We have previously reported on alternative methods of evaluating HRQL, solutions for missing data in clinical trials as well as tested statistical and clinically meaningful differences, within and between treatment groups, in clinical trials with patients diagnosed with hepatobiliary carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with HCC seen at UPMC will be enrolled in this study if they meet the following eligibility criteria:
* Adults patients (≥ 18 years of age) with a diagnosis of HCC which is not amenable to surgical resection or local ablative therapy
* Histological confirmed HCC or clinical/laboratory diagnosis of HCC or nodules larger than 2 cm with typical vascular features or AFP > 200
* Patient must have quantifiable disease limited to the liver
* Patients must have at least one tumor lesion that meets both of the following criteria:

  * The lesion can be accurately measured in at least one dimension according to RECIST criteria
  * The lesion has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* ECOG performance status (PS) <2
* No prior targeted antiangiogenic therapy. Metronomic chemotherapies are allowed. At least 4 weeks since prior systemic chemotherapy
* At least 4 weeks since prior TACE
* At least 4 weeks since prior interferon
* Not pregnant
* No significant baseline liver dysfunction. Cirrhotic status of Child-Pugh class A only
* No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
* No current infections requiring antibiotic therapy
* Not on anticoagulation or suffering from a known bleeding disorder
* No unstable coronary artery disease or recent MI
* The following laboratory parameters:

  * Platelet count ≥ 60,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or a Pt/PTT within normal limits
  * Absolute neutrophil count (ANC) > 1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC except cervical carcinoma in situ, treated basal-cell carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), and any cancer curatively treated > 3 years prior to entry is permitted
* Renal failure requiring hemo- or peritoneal dialysis
* Child-Pugh B & C hepatic impairment
* History of cardiac disease: > NY Heart Association (NYHA) class 2 congestive heart failure, active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, and uncontrolled hypertension. Myocardial infarction more than 6 months prior to study entry is permitted.
* Active clinically serious infections (> CTCAEv3 grade 2)
* Known history of HIV
* Known central nervous system tumors including metastatic brain disease
* History of organ allograft
* Substance abuse (current), psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Patients unable to swallow oral medications.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of the study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg, despite optimal medical management
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture

Excluded therapies and medications, previous and concomitant:

* Prior use of Raf-kinase inhibitors (RKI), VEGF inhibitors, MEK inhibitors, or farnesyl transferase inhibitors
* Major surgery within 6 weeks of start of study drug
* Radiotherapy during study or within 3 weeks prior to start of study drug.
* Use of biologic response modifiers such as granulocyte colony-stimulating factor (G-CSF) within 3 weeks prior to study entry.
* Autologous bone marrow transplant or stem cell rescue within four months of study drug initiation
* Concomitant treatment with rifampin or St. John's wort.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Gamblin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tace + Sorafenib: Patients with unresectable HCC will be treated with TACE in combination with oral sorafenib administration. TACE will be accomplished with gelatin microspheres (Embospheres) following delivery of 125 mg/m2 of cisplatin. Oral sorafenib (400 mg BID) will start the next day after the first TACE treatment.
  TACE + Sorafenib: TACE will be accomplished with gelatin microspheres (Embospheres) following delivery of 125 mg/m2 of cisplatin. Oral sorafenib (400 mg BID) will start the next day after the first TACE treatment until unacceptable toxicity occurs, or until study termination.
Period: Overall Study
Arm/Group | Tace + Sorafenib
Started | 19
Completed | 5
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 2
Not completed — did not meet eligibility criteria | 8
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tace + Sorafenib
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 11
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Determine Progression-free Survival in This Patient Population Treated With the Proposed Combination Treatment Modality
Description: Progression free survival (PFS) is calculated as the time interval between the date on which a patient first received protocol treatment and the documented date of disease progression or death. For a surviving and progression-free patient, PFS is censored by the last follow-up date when that patient is documented to be progression free. Progression is defined using RECIST v1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measureable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 24 months (from initial treatment through 12 months follow-up)
Population: Patients who received at least one cycle of the entire treatment regimen (this did not include two patients who went on to receive liver transplants).
Measure: Median (Full Range); unit: days
Arm/Group | Tace + Sorafenib
Number analyzed (Participants) | 6
days | 174.00 [.000 to 427.355]

2. Secondary Outcome: Determine the Overall Survival in Patients Treated With This Combination Regimen
Description: Overall survival (OS) is calculated as the time interval between the date on which a patient first received protocol treatment and the documented date of death. For a surviving patient, OS is censored by the last follow-up date when that patient is documented to be alive.
Time Frame: From date of initial treatment until the date of death from any cause
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Tace + Sorafenib
Number analyzed (Participants) | 6
days | 156.000 [.000 to 991.374]

ADVERSE EVENTS:
Description: Regular investigator assessment and laboratory testing in addition to participant self reporting
Arm/Group | Tace + Sorafenib
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tace + Sorafenib (N=19)
renal failure (Renal and urinary disorders) | 1 (1) — The PI determined that this event was possibly related to TACE/nexavar intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tace + Sorafenib (N=19)
Increased ALT (Investigations) | 4 (4)
Increased AST (Blood and lymphatic system disorders) | 5 (5)
Fatigue (General disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 3 (3)
Increased GGTP (Investigations) | 5 (5)
leukopenia (Investigations) | 3 (3)
thrombocytopenia (Investigations) | 4 (4)
Increased total bilirubin (Investigations) | 5 (5)
nausea (Gastrointestinal disorders) | 1 (1)
Hiccups (General disorders) | 2 (2)
Increased Alkaline Phosphatase (Investigations) | 2 (2)
Hypophosphatemia (Investigations) | 2 (2)
Increased Lipase (Investigations) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hoarseness (General disorders) | 5 (5)
Abdominal Pain (General disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Tremors (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Weight Loss (Investigations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Mouth Infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Decreased Serum Albumin (Metabolism and nutrition disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Bloating (Gastrointestinal disorders) | 2 (2)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Breast Tenderness (Reproductive system and breast disorders) | 1 (1)
Bleeding oral cavity (Gastrointestinal disorders) | 1 (1)
Increased urination (Renal and urinary disorders) | 1 (1)
Difficulty swallowing (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Bleeding varices (Gastrointestinal disorders) | 1 (1)
Lower Extremity Edema (General disorders) | 1 (1)
Incisional hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 1 (1)
Elevated Amylase (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No